CLINICAL TRIAL: NCT01999335
Title: Phase 1b/3 Multicenter Study of Oprozomib, Pomalidomide, and Dexamethasone in Primary Refractory or Relapsed and Refractory Multiple Myeloma Subjects
Brief Title: A Study of Oprozomib, Pomalidomide, and Dexamethasone in Adults With Primary Refractory or Relapsed and Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: A program evaluation identified that the safety profile and pharmacokinetic (PK) characteristics of the formulation used in all oprozomib studies required further optimization and thus enrollment in OPZ007 was halted during dose-expansion.
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: OPZ007; 20130411 (Other: Amgen Study ID)
Record Dates: First submitted 2013-11-25; First posted 2013-12-03 (Estimated); Results first posted 2021-04-27 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-03

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — ONX 0912; pomalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Oprozomib 150 mg 5/14 + Pomalidomide 4 mg + Dexamethasone (Experimental): Participants received oprozomib 150 mg once daily on days 1 to 5 and days 15 to 19 (5/14 schedule) of each 28-day treatment cycle, in combination with pomalidomide 4 mg/day on days 1 to 21 and dexamethasone 20 mg on days 1, 2, 8, 9, 15, 16, 22, and 23 of each 28-day cycle until disease progression or unacceptable toxicity.
  Interventions: Drug: Oprozomib; Drug: Pomalidomide; Drug: Dexamethasone
- Oprozomib 150 mg 5/14 + Pomalidomide 2 mg + Dexamethasone (Experimental): Participants received oprozomib 150 mg once daily on days 1 to 5 and days 15 to 19 (5/14 schedule) of each 28-day treatment cycle, in combination with pomalidomide 2 mg/day on days 1 to 21 and dexamethasone 20 mg on days 1, 2, 8, 9, 15, 16, 22, and 23 of each 28-day cycle until disease progression or unacceptable toxicity.
  Interventions: Drug: Oprozomib; Drug: Pomalidomide; Drug: Dexamethasone
- Oprozomib 210 mg 2/7 + Pomalidomide 4 mg + Dexamethasone (Experimental): Participants received oprozomib 210 mg once daily on days 1, 2, 8, 9, 15, 16, 22, and 23 (2/7 schedule) of each 28-day treatment cycle, in combination with pomalidomide 4 mg on days 1 through 21 and dexamethasone 20 mg/day on days 1, 2, 8, 9, 15, 16, 22, and 23 of each 28-day cycle until disease progression or unacceptable toxicity.
  Interventions: Drug: Oprozomib; Drug: Pomalidomide; Drug: Dexamethasone
- Oprozomib 240 mg 2/7 + Pomalidomide 4 mg + Dexamethasone (Experimental): Participants received oprozomib 240 mg once daily on days 1, 2, 8, 9, 15, 16, 22, and 23 (2/7 schedule) of each 28-day treatment cycle, in combination with pomalidomide 4 mg on days 1 through 21 and dexamethasone 20 mg/day on days 1, 2, 8, 9, 15, 16, 22, and 23 of each 28-day cycle until disease progression or unacceptable toxicity.
  Interventions: Drug: Oprozomib; Drug: Pomalidomide; Drug: Dexamethasone
- Oprozomib 210 mg 2/7 + Pomalidomide 4 mg + Dexamethasone: Expansion Phase (Experimental): Participants received oprozomib 210 mg once daily on days 1, 2, 8, 9, 15, 16, 22, and 23 (2/7 schedule) of each 28-day treatment cycle, in combination with pomalidomide 4 mg on days 1 through 21 and dexamethasone 20 mg/day on days 1, 2, 8, 9, 15, 16, 22, and 23 of each 28-day cycle until disease progression or unacceptable toxicity.
  Interventions: Drug: Oprozomib; Drug: Pomalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Oprozomib — Extended release (ER) tablets administered orally
Drug: Pomalidomide — Capsules for oral administration
  Other Names: POMALYST®
Drug: Dexamethasone — Tablets for oral administration

SUMMARY:
The purpose of the Phase 1 part of the study is to determine the maximum tolerated dose and assess the safety, tolerability and activity of oprozomib in combination with pomalidomide and dexamethasone in adults with primary refractory or relapsed and refractory multiple myeloma.

The purpose of the Phase 3 part of the study is to compare the efficacy for adults with primary refractory or relapsed and refractory multiple myeloma who are randomized to either oprozomib or placebo in combination with pomalidomide and dexamethasone.

DETAILED DESCRIPTION:
This was a phase 1b/3, multicenter study composed of 2 parts: part 1 was a phase 1b, open-label, dose-escalation and dose-expansion component and part 2 was to have been a phase 3, placebo-controlled, double-blind, randomized component. Part 2 was not conducted.

The Phase 1 dose-escalation portion of the study followed a standard 3 + 3 dose-escalation design. For each of the 2 schedules, groups of 3 to 6 patients were enrolled. The starting doses of oprozomib were 150 and 210 mg in the 5/14 and 2/7 schedules, respectively. The starting dose of pomalidomide was 4 mg in both schedules. As long as < 33% of patients experienced a dose-limiting toxicity (DLT) in a given cohort, the dose of oprozomib was escalated in 30-mg increments for successive cohorts.

Once the recommended dose and schedule for the expansion phase had been selected, additional participants were enrolled in the dose expansion portion of part 1 to continue the evaluation of the safety and efficacy of the regimen and determine the recommended phase 3 dose. Enrollment was halted during the dose expansion phase and part 2 was not conducted.

ELIGIBILITY:
Key Inclusion Criteria:

1. Multiple myeloma that is primary refractory or relapsed and refractory after at least 2 lines of standard for multiple myeloma including:

   1. ≥ 2 consecutive cycles of both bortezomib and lenalidomide or thalidomide (alone or in combination)
   2. In the dose-expansion and Phase 3 portions of the study only: In addition to the above, treatment with adequate alkylator therapy, defined as:

   i. High-dose melphalan or other alkylating agent as conditioning for autologous or allogeneic stem cell transplant (SCT), or ii. ≥ 6 cycles of induction therapy, or iii. Progressive disease after ≥ 2 cycles
2. Disease progression on or within 60 days of completion of the last therapy
3. Measurable disease as indicated by 1 or more of the following:

   1. Serum M-protein ≥ 500 mg/dL
   2. Urine M-protein ≥ 200 mg/24 h
   3. For patients without measurable serum or urine M protein, serum free light chain (SFLC): Involved free light chain (FLC) concentration ≥ 10 mg/dL provided SFLC ratio is abnormal
4. Males and females ≥ 18 years old
5. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2

Key Exclusion Criteria:

1. Systemic chemotherapy with approved or investigational anticancer therapeutics, intended to treat underlying malignancy, within 3 weeks before the first dose or 6 weeks for antibody therapy
2. Dexamethasone at cumulative doses greater than 160 mg or equivalent within 21 days prior to the first dose of study treatment is not allowed. Use of topical or inhaled steroids is acceptable.
3. Radiation therapy within 3 weeks before first dose. Radioimmunotherapy within 8 weeks before first dose.
4. Plasmapheresis is not permitted at any time during the Screening period or while the subject is receiving study treatment. If a subject has started Screening procedures requiring plasmapheresis, or is anticipated to require plasmapheresis during or after the Screen
5. Autologous SCT within 8 weeks or allogeneic SCT within 16 weeks prior to initiation of study treatment. Patients with prior allogeneic SCT should not have evidence of moderate-to-severe graft-versus-host disease (as defined in Filipovich 2005).
6. Known hypersensitivity to any immunomodulatory drugs (IMiDs), including Grade 4 rash
7. Prior treatment of any duration with pomalidomide
8. Known hypersensitivity or intolerance to dexamethasone
9. Prior exposure to oprozomib
10. Congestive heart failure (New York Heart Association Class III to IV), symptomatic ischemia, conduction abnormalities uncontrolled by conventional intervention, or myocardial infarction within 6 months before first dose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2014-07-30 (Actual); Primary Completion 2019-04-25 (Actual); Study Completion 2019-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (17):
- United States (17):
  - California Cancer Associates For Research and Exellence, cCare, Encinitas, California
  - James R. Berenson, MD, Inc., West Hollywood, California
  - Innovative Clinical Research Institute, Whittier, California
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Oncology Hematology West PC, dba Nebraska Cancer Specialists, Omaha, Nebraska
  - Weill Cornell Medical College-New York Presbyterian Hospital, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Willamette Valley Cancer Institute and Research Center, Springfield, Oregon
  - Abramson Cancer Center of the University of Pennsylvania at Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Tennessee Oncology, PLLC / Sarah Cannon Research Institute, Nashville, Tennessee
  - The University of Texas M.D. Anderson Cancer Center, Houston, Texas
  - Cancer Care Centers of South Texas-HOAST, San Antonio, Texas
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Yakima Valley Memorial Hospital/North Star Lodge, Yakima, Washington

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 12 centers in the United States. This study was composed of 2 parts: part 1 was a phase 1b, open-label, dose-escalation and dose-expansion component and part 2 was to have been a phase 3, placebo-controlled, double-blind, randomized component. Part 2 was not conducted.
Pre-assignment Details: In part 1 participants were enrolled sequentially using a standard 3 + 3 dose escalation schema. Additional participants were to be enrolled in the dose expansion portion once the recommended dose and schedule had been selected; enrollment was halted after 12 participants were enrolled in the expansion cohort.
Period: Overall Study
Arm/Group | Oprozomib 150 mg 5/14 + Pomalidomide 4 mg + Dexamethasone | Oprozomib 150 mg 5/14 + Pomalidomide 2 mg + Dexamethasone | Oprozomib 210 mg 2/7 + Pomalidomide 4 mg + Dexamethasone | Oprozomib 240 mg 2/7 + Pomalidomide 4 mg + Dexamethasone | Oprozomib 210 mg 2/7 + Pomalidomide 4 mg + Dexamethasone: Expansion Phase
Started | 3 | 1 | 7 | 10 | 12
Received Study Treatment | 3 | 1 | 7 | 10 | 10
Completed | 3 | 1 | 7 | 10 | 10
Not Completed | 0 | 0 | 0 | 0 | 2
Not completed — Discontinued before receiving treatment | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: The safety population included all participants who received at least 1 dose of any study treatment
Groups:
- Total: Total of all reporting groups
Arm/Group | Oprozomib 150 mg 5/14 + Pomalidomide 4 mg + Dexamethasone | Oprozomib 150 mg 5/14 + Pomalidomide 2 mg + Dexamethasone | Oprozomib 210 mg 2/7 + Pomalidomide 4 mg + Dexamethasone | Oprozomib 240 mg 2/7 + Pomalidomide 4 mg + Dexamethasone | Oprozomib 210 mg 2/7 + Pomalidomide 4 mg + Dexamethasone: Expansion Phase | Total
Number analyzed (Participants) | 3 | 1 | 7 | 10 | 10 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.7 (5.5) | 59.0 | 57.1 (12.9) | 68.2 (7.3) | 63.7 (6.0) | 62.6 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 3 | 2 | 5 | 13
  Male | 0 | 1 | 4 | 8 | 5 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 2 | 1 | 0 | 3
  Not Hispanic or Latino | 3 | 1 | 4 | 8 | 8 | 24
  Unknown or Not Reported | 0 | 0 | 1 | 1 | 2 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Black | 1 | 0 | 2 | 4 | 1 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  White | 2 | 1 | 4 | 6 | 7 | 20
  Not reported | 0 | 0 | 1 | 0 | 2 | 3
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — A scale to assess a patient's disease status. 0 = Fully active, able to carry out all pre-disease performance without restriction;
  1. = Restricted in physically strenuous activity, ambulatory and able to carry out work of a light nature;
  2. = Ambulatory and capable of all self-care, unable to carry out any work activities. Up and about > 50% of waking hours;
  3. = Capable of only limited self-care, confined to bed or chair > 50% of waking hours;
  4. = Completely disabled, confined to bed or chair;
  5. = Dead.
  Participants
    Grade 0 (Fully active) | 0 | 0 | 2 | 4 | 3 | 9
    Grade 1 (Restricted but ambulatory) | 3 | 1 | 5 | 4 | 6 | 19
    Grade 2 (Ambulatory but unable to work) | 0 | 0 | 0 | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-limiting Toxicities (DLTs)
Description: DLTs were assessed according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.03, defined as any of the following treatment-related events occurring within 4 weeks after the first dose of therapy:
  Any grade ≥ 3 nonhematologic toxicity, except: Grade 3 asymptomatic electrolyte abnormalities or hypophosphatemia for < 24 hours; Grade 3 nausea, vomiting or diarrhea unless for > 3 days despite optimal supportive care; Grade 3 fatigue for < 14 days; Grade ≥ 3 hyperglycemia or toxicity attributed to dexamethasone and Grade ≥ 3 rash attributed to pomalidomide.
  Hematologic toxicities:
  * Grade 4 neutropenia: Absolute neutrophil count < 0.5 × 10^9/L for ≥ 7 days despite adequate growth factor support; febrile neutropenia
  * Thrombocytopenia: Grade 4 for ≥ 7 days, or Grade 4 for < 7 days with grade 2 clinically significant bleeding or < 10,000 platelets requiring transfusion, or Grade 3 with clinically significant bleeding or requiring platelet transfusion.
Time Frame: Cycle 1, 28 days
Population: Participants who received at least 1 dose of any study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Oprozomib 150 mg 5/14 + Pomalidomide 4 mg + Dexamethasone | Oprozomib 150 mg 5/14 + Pomalidomide 2 mg + Dexamethasone | Oprozomib 210 mg 2/7 + Pomalidomide 4 mg + Dexamethasone | Oprozomib 240 mg 2/7 + Pomalidomide 4 mg + Dexamethasone | Oprozomib 210 mg 2/7 + Pomalidomide 4 mg + Dexamethasone: Expansion Phase
Number analyzed (Participants) | 3 | 1 | 7 | 10 | 10
Participants
  Any dose-limiting toxicity | 2 | 0 | 1 | 0 | 0
  Gastric hemorrhage | 0 | 0 | 1 | 0 | 0
  Abdominal distension | 1 | 0 | 0 | 0 | 0
  Cognitive disorder | 1 | 0 | 0 | 0 | 0
  Mucosal inflammation | 1 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: Adverse events (AEs) were graded using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.03 and according to the following: Grade 1 = mild AE, Grade 2 = Moderate AE, Grade 3 = a severe AE, Grade 4 = life-threatening AE, and Grade 5 = death due to AE.
  A serious AE is an event that met 1 or more of the following criteria:
  * Death
  * Life-threatening experience
  * Required inpatient hospitalization or prolongation of an existing hospitalization
  * Resulted in persistent or significant disability/incapacity
  * A congenital anomaly birth defect in the offspring of an exposed female subject or offspring of a female partner of a male subject
  * Important medical events that, based upon appropriate medical judgment, jeopardized the participant and may have required medical or surgical intervention to prevent an outcome listed above.
  Treatment-related AEs (TRAE) are those considered related to at least 1 study drug by the investigator.
Time Frame: From first dose of any study drug up to 30 days after the last dose; median duration of treatment was 7.6, 28.0, 32.1, 46.3, and 17.4 weeks in each treatment group, respectively.
Population: Participants who received at least 1 dose of any study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Oprozomib 150 mg 5/14 + Pomalidomide 4 mg + Dexamethasone | Oprozomib 150 mg 5/14 + Pomalidomide 2 mg + Dexamethasone | Oprozomib 210 mg 2/7 + Pomalidomide 4 mg + Dexamethasone | Oprozomib 240 mg 2/7 + Pomalidomide 4 mg + Dexamethasone | Oprozomib 210 mg 2/7 + Pomalidomide 4 mg + Dexamethasone: Expansion Phase
Number analyzed (Participants) | 3 | 1 | 7 | 10 | 10
Participants
  Any treatment-emergent adverse event | 3 | 1 | 7 | 10 | 10
  TEAE Grade ≥ 3 | 2 | 1 | 5 | 9 | 9
  Serious adverse events | 0 | 1 | 3 | 6 | 6
  TEAEs leading to discontinuation of study drug | 1 | 0 | 2 | 1 | 4
  Fatal adverse events | 0 | 0 | 0 | 0 | 0
  Treatment-related treatment-emergent adverse events (TRAE) | 3 | 1 | 7 | 10 | 10
  Treatment-related TEAE Grade ≥ 3 | 2 | 1 | 4 | 6 | 7
  Treatment-related serious adverse events | 0 | 0 | 1 | 2 | 2
  TRAEs leading to discontinuation of study drug | 1 | 0 | 1 | 1 | 4
  Treatment-related fatal adverse events | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as the percentage of participants with a best overall response of partial response (PR), very good PR (VGPR), complete response (CR), or stringent CR (sCR) based on the International Myeloma Working Group Uniform Response Criteria.
  PR: ≥ 50% reduction of serum M-protein and ≥90% reduction in urine M-protein or to < 200 mg/24 hrs, or a ≥50% decrease in the difference between involved and uninvolved free light chain levels (dFLC). A ≥ 50% decrease in the size of soft tissue plasmacytomas present at baseline.
  VGPR: Serum and urine M-protein detectable by immunofixation but not electrophoresis or ≥ 90% decrease in serum M-protein with urine M-protein <100 mg/24 hrs. If disease measurable only by serum FLC (SFLC), ≥ 90% decrease in dFLC.
  CR: No immunofixation on serum and urine, disappearance of soft tissue plasmacytomas and <5% plasma cells in bone marrow (BM). Normal SFLC ratio if disease measurable only by SFLC.
  sCR: As for CR, and absence of clonal plasma cells in BM.
Time Frame: Disease response was assessed every 4 weeks for the first 18 months and then every 8 weeks for the remainder of study treatment; median duration of treatment was 7.6, 28.0, 32.1, 46.3, and 17.4 weeks in each treatment group, respectively.
Population: Participants who received at least 1 dose of any study drug
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Oprozomib 150 mg 5/14 + Pomalidomide 4 mg + Dexamethasone | Oprozomib 150 mg 5/14 + Pomalidomide 2 mg + Dexamethasone | Oprozomib 210 mg 2/7 + Pomalidomide 4 mg + Dexamethasone | Oprozomib 240 mg 2/7 + Pomalidomide 4 mg + Dexamethasone | Oprozomib 210 mg 2/7 + Pomalidomide 4 mg + Dexamethasone: Expansion Phase
Number analyzed (Participants) | 3 | 1 | 7 | 10 | 10
percentage of participants | 33.3 [0.8 to 90.6] | 100.0 [2.5 to 100.0] | 85.7 [42.1 to 99.6] | 60.0 [26.2 to 87.8] | 60.0 [26.2 to 87.8]

4. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: Clinical benefit rate is defined as the percentage of participants with a best overall response of minimal response (MR) per modified European Group for Blood and Marrow Transplantation criteria, or PR, VGPR, CR, or sCR as determined by the investigator according to the International Myeloma Working Group Uniform Response Criteria (IMWG-URC).
  MR:
  * ≥ 25% but < 49% reduction in serum M-protein and a 50 - 89% reduction in 24-hour urinary M-protein, which still exceeds 200 mg per 24 hours
  * If the serum and urine M-protein were not measurable, a decrease of 25 - 49% in the difference between involved and uninvolved FLC levels was required in place of the M-protein criteria.
  * For patients with nonsecretory myeloma only, 25 - 49% reduction in plasma cells in a bone marrow aspirate and on trephine biopsy, if biopsy is performed
  * 25 - 49% reduction in the size of soft tissue plasmacytomas (by radiography or clinical examination)
Time Frame: as for outcome 3
Population: Participants who received at least 1 dose of any study drug
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Oprozomib 150 mg 5/14 + Pomalidomide 4 mg + Dexamethasone | Oprozomib 150 mg 5/14 + Pomalidomide 2 mg + Dexamethasone | Oprozomib 210 mg 2/7 + Pomalidomide 4 mg + Dexamethasone | Oprozomib 240 mg 2/7 + Pomalidomide 4 mg + Dexamethasone | Oprozomib 210 mg 2/7 + Pomalidomide 4 mg + Dexamethasone: Expansion Phase
Number analyzed (Participants) | 3 | 1 | 7 | 10 | 10
percentage of participants | 33.3 [0.8 to 90.6] | 100.0 [2.5 to 100.0] | 85.7 [42.1 to 99.6] | 60.0 [26.2 to 87.8] | 60.0 [26.2 to 87.8]

5. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Oprozomib
Description: Oprozomib plasma concentrations were determined using liquid chromatography with tandem mass spectrometry.
Time Frame: Cycle 1 day 1 at predose and 0.25, 0.5, 1, 2, 3, 4, 6, and 24 hours postdose. Cycle 2 day 1 at predose and 0.25, 0.5, 1, 2, 3, 4, and 6 hours postdose.
Population: Participants with adequate oprozomib plasma concentration-versus-time data to allow estimation of pharmacokinetic (PK) parameters. Treatment groups receiving the same dose of oprozomib were combined for PK analyses.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Oprozomib 150 mg 5/14 + Pomalidomide + Dexamethasone: Participants received oprozomib 150 mg once daily on days 1 to 5 and days 15 to 19 (5/14 schedule) of each 28-day treatment cycle, in combination with pomalidomide 2 or 4 mg/day on days 1 to 21 and dexamethasone 20 mg on days 1, 2, 8, 9, 15, 16, 22, and 23 of each 28-day cycle.
- Oprozomib 210 mg 2/7 + Pomalidomide + Dexamethasone: Participants received oprozomib 210 mg once daily on days 1, 2, 8, 9, 15, 16, 22, and 23 (2/7 schedule) of each 28-day treatment cycle, in combination with pomalidomide 4 mg on days 1 through 21 and dexamethasone 20 mg/day on days 1, 2, 8, 9, 15, 16, 22, and 23 of each 28-day cycle.
Arm/Group | Oprozomib 150 mg 5/14 + Pomalidomide + Dexamethasone | Oprozomib 210 mg 2/7 + Pomalidomide + Dexamethasone | Oprozomib 240 mg 2/7 + Pomalidomide 4 mg + Dexamethasone
Number analyzed (Participants) | 3 | 16 | 9
ng/mL
  Cycle 1 day 1 | 492 (398.3) | 744 (119.4) | 757 (38.7)
  Cycle 2 day 1: number analyzed (Participants) | 3 | 14 | 7
  Cycle 2 day 1 | 181 (401.1) | 1030 (91.5) | 965 (44.4)

6. Primary Outcome: Number of Participants With Post-Baseline Grade 3 or 4 Laboratory Toxicities
Description: Laboratory abnormalities were graded using National Cancer Institute Common Terminology Criteria for Adverse Events (version 4.03).
  Full chemistry panel included sodium, potassium, calcium, alkaline phosphatase, blood urea nitrogen, uric acid, lactate dehydrogenase, creatinine, chloride, bicarbonate, glucose, total protein, albumin, total bilirubin, alanine aminotransferase (ALT), aspartate aminotransferase (AST), phosphorous, and magnesium.
  Complete blood count (CBC) with differential included hemoglobin, hematocrit, white blood cell (WBC) count with complete manual or automated differential (total neutrophils, lymphocytes, monocytes, eosinophils, basophils; reported as absolute counts), red blood cell (RBC) count, and platelet count.
Time Frame: Cycles 1 and 2 days 1, 5, 15, and 19 and days 3 and 8 of cycle 1, and day 1 of each cycle from cycle 3 thereafter until the end of treatment; median duration of treatment was 7.6, 28.0, 32.1, 46.3, and 17.4 weeks in each treatment group, respectively.
Population: Participants who received at least 1 dose of any study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Oprozomib 150 mg 5/14 + Pomalidomide 4 mg + Dexamethasone | Oprozomib 150 mg 5/14 + Pomalidomide 2 mg + Dexamethasone | Oprozomib 210 mg 2/7 + Pomalidomide 4 mg + Dexamethasone | Oprozomib 240 mg 2/7 + Pomalidomide 4 mg + Dexamethasone | Oprozomib 210 mg 2/7 + Pomalidomide 4 mg + Dexamethasone: Expansion Phase
Number analyzed (Participants) | 3 | 1 | 7 | 10 | 10
Participants
  At least 1 Grade 3 or 4 laboratory toxicity | 2 | 1 | 6 | 8 | 8
  Grade 3 increase in glucose | 0 | 0 | 0 | 1 | 1
  Grade 4 increase in glucose | 0 | 0 | 0 | 1 | 0
  Grade 3 increase in total bilirubin | 0 | 0 | 0 | 1 | 0
  Grade 3 increase in magnesium | 0 | 0 | 0 | 0 | 1
  Grade 4 decrease in magnesium | 0 | 0 | 0 | 1 | 0
  Grade 3 decrease in sodium | 0 | 0 | 0 | 3 | 0
  Grade 4 decrease in sodium | 0 | 0 | 0 | 1 | 0
  Grade 3 decrease in hemoglobin | 1 | 1 | 2 | 1 | 3
  Grade 3 decrease in leukocytes | 1 | 1 | 1 | 1 | 2
  Grade 4 decrease in leukocytes | 0 | 0 | 0 | 0 | 1
  Grade 3 decrease in neutrophils | 2 | 1 | 3 | 1 | 4
  Grade 4 decrease in neutrophils | 0 | 0 | 0 | 0 | 2
  Grade 3 decrease in lymphocytes | 1 | 0 | 5 | 3 | 4
  Grade 4 decrease in lymphocytes | 0 | 0 | 0 | 2 | 0
  Grade 3 decrease in platelets | 1 | 0 | 0 | 2 | 5

7. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of Oprozomib
Description: Oprozomib plasma concentrations were determined using liquid chromatography with tandem mass spectrometry.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Median (Full Range); unit: hours
Arm/Group | Oprozomib 150 mg 5/14 + Pomalidomide + Dexamethasone | Oprozomib 210 mg 2/7 + Pomalidomide + Dexamethasone | Oprozomib 240 mg 2/7 + Pomalidomide 4 mg + Dexamethasone
Number analyzed (Participants) | 3 | 16 | 9
hours
  Cycle 1 day 1 | 1.0 [1.0 to 6.1] | 1.6 [0.5 to 6.1] | 2.2 [1.1 to 3.8]
  Cycle 2 day 1: number analyzed (Participants) | 3 | 14 | 7
  Cycle 2 day 1 | 4.0 [1.0 to 4.1] | 1.1 [0.42 to 4.0] | 1.1 [0.63 to 4.0]

8. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to Time of Last Quantifiable Concentration (AUClast) of Oprozomib
Description: Oprozomib plasma concentrations were determined using liquid chromatography with tandem mass spectrometry.
  The area under the plasma concentration-time curve from time 0 to time of last quantifiable concentration (AUClast) was estimated using the linear trapezoidal method.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Oprozomib 150 mg 5/14 + Pomalidomide + Dexamethasone | Oprozomib 210 mg 2/7 + Pomalidomide + Dexamethasone | Oprozomib 240 mg 2/7 + Pomalidomide 4 mg + Dexamethasone
Number analyzed (Participants) | 3 | 16 | 9
hr*ng/mL
  Cycle 1 day 1 | 1090 (192.2) | 1700 (145.9) | 1730 (48.7)
  Cycle 2 day 1: number analyzed (Participants) | 3 | 14 | 7
  Cycle 2 day 1 | 446 (605.7) | 1860 (81.9) | 1800 (17.2)

9. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to Time Infinity (AUCinf) of Oprozomib
Description: Oprozomib plasma concentrations were determined using liquid chromatography with tandem mass spectrometry.
  The area under the plasma concentration-time curve from time 0 to time infinity (AUCinf), estimated as the sum of AUClast and Clast/λz, where Clast is the last predicted concentration and λz is the first-order terminal rate constant estimated via linear regression of the terminal log-linear decay phase.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Oprozomib 150 mg 5/14 + Pomalidomide + Dexamethasone | Oprozomib 210 mg 2/7 + Pomalidomide + Dexamethasone | Oprozomib 240 mg 2/7 + Pomalidomide 4 mg + Dexamethasone
Number analyzed (Participants) | 2 | 8 | 5
hr*ng/mL
  Cycle 1 day 1: number analyzed (Participants) | 2 | 5 | 4
  Cycle 1 day 1 | 2250 (NA) — Not calculated when N ≤ 2 | 3440 (96.1) | 1660 (35.8)
  Cycle 2 day 1: number analyzed (Participants) | 0 | 8 | 5
  Cycle 2 day 1 |  | 1830 (87.7) | 1900 (12.4)

ADVERSE EVENTS:
Time Frame: All-cause mortality: From the date of enrollment until the data cutoff of 25 April 2019, a maximum of 51 months. Treatment-emergent adverse events: From the first dose of any study treatment and within the end of study or 30 days of the last dose of any study treatment, whichever occurred earlier; median duration of treatment was 7.6, 28.0, 32.1, 46.3, and 17.4 weeks in each treatment group, respectively.
Description: All-cause mortality is reported for all participants enrolled in the study. Serious adverse events and other adverse events are reported for all participants who received at least one dose of any study drug.
Arm/Group | Oprozomib 150 mg 5/14 + Pomalidomide 4 mg + Dexamethasone | Oprozomib 150 mg 5/14 + Pomalidomide 2 mg + Dexamethasone | Oprozomib 210 mg 2/7 + Pomalidomide 4 mg + Dexamethasone | Oprozomib 240 mg 2/7 + Pomalidomide 4 mg + Dexamethasone | Oprozomib 210 mg 2/7 + Pomalidomide 4 mg + Dexamethasone: Expansion Phase
All-Cause Mortality (participants affected / at risk) | 1/3 | 0/1 | 4/7 | 3/10 | 4/12
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/1 | 3/7 | 6/10 | 6/10
Other Adverse Events (participants affected / at risk) | 3/3 | 1/1 | 7/7 | 10/10 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oprozomib 150 mg 5/14 + Pomalidomide 4 mg + Dexamethasone (N=3) | Oprozomib 150 mg 5/14 + Pomalidomide 2 mg + Dexamethasone (N=1) | Oprozomib 210 mg 2/7 + Pomalidomide 4 mg + Dexamethasone (N=7) | Oprozomib 240 mg 2/7 + Pomalidomide 4 mg + Dexamethasone (N=10) | Oprozomib 210 mg 2/7 + Pomalidomide 4 mg + Dexamethasone: Expansion Phase (N=10)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 3
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
GASTRIC HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
PYREXIA (General disorders) | 0 | 0 | 0 | 0 | 1
ABSCESS JAW (Infections and infestations) | 0 | 0 | 0 | 1 | 0
CELLULITIS (Infections and infestations) | 0 | 0 | 1 | 0 | 0
INFLUENZA (Infections and infestations) | 0 | 1 | 0 | 1 | 0
ORAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 1 | 0
PARAINFLUENZAE VIRUS INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 1
PLEURAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 1 | 0
PNEUMONIA (Infections and infestations) | 0 | 1 | 0 | 2 | 2
PNEUMONIA VIRAL (Infections and infestations) | 0 | 0 | 0 | 0 | 1
SEPSIS (Infections and infestations) | 0 | 0 | 1 | 0 | 0
SINUSITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 1
VIRAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 1 | 0
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
RIB FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
NEUTROPHIL COUNT DECREASED (Investigations) | 0 | 0 | 0 | 0 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
COGNITIVE DISORDER (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
HAEMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Oprozomib 150 mg 5/14 + Pomalidomide 4 mg + Dexamethasone (N=3) | Oprozomib 150 mg 5/14 + Pomalidomide 2 mg + Dexamethasone (N=1) | Oprozomib 210 mg 2/7 + Pomalidomide 4 mg + Dexamethasone (N=7) | Oprozomib 240 mg 2/7 + Pomalidomide 4 mg + Dexamethasone (N=10) | Oprozomib 210 mg 2/7 + Pomalidomide 4 mg + Dexamethasone: Expansion Phase (N=10)
ANAEMIA (Blood and lymphatic system disorders) | 1 | 1 | 3 | 4 | 7
HYPERCOAGULATION (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
INCREASED TENDENCY TO BRUISE (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
LEUKOPENIA (Blood and lymphatic system disorders) | 0 | 1 | 1 | 1 | 3
NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 1 | 3 | 2 | 3
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 | 1 | 1 | 1 | 6
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
PALPITATIONS (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
TACHYCARDIA (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
TINNITUS (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
VERTIGO (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 2
CATARACT (Eye disorders) | 0 | 0 | 1 | 0 | 1
DRY EYE (Eye disorders) | 0 | 0 | 1 | 0 | 2
EYE HAEMATOMA (Eye disorders) | 0 | 0 | 0 | 1 | 0
EYE IRRITATION (Eye disorders) | 0 | 0 | 1 | 0 | 0
LACRIMATION INCREASED (Eye disorders) | 0 | 0 | 0 | 0 | 1
PERIORBITAL OEDEMA (Eye disorders) | 0 | 1 | 0 | 0 | 0
SCLERAL HAEMORRHAGE (Eye disorders) | 0 | 0 | 0 | 1 | 0
VISION BLURRED (Eye disorders) | 1 | 0 | 0 | 1 | 2
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 | 0 | 2 | 4 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2
CONSTIPATION (Gastrointestinal disorders) | 2 | 0 | 3 | 6 | 6
DENTAL DISCOMFORT (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
DIARRHOEA (Gastrointestinal disorders) | 2 | 0 | 7 | 9 | 8
DIVERTICULAR PERFORATION (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
DYSPEPSIA (Gastrointestinal disorders) | 1 | 0 | 3 | 3 | 3
ERUCTATION (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
FLATULENCE (Gastrointestinal disorders) | 1 | 0 | 2 | 3 | 0
FREQUENT BOWEL MOVEMENTS (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
GASTROINTESTINAL PAIN (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 1
GINGIVAL PAIN (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
HYPOAESTHESIA ORAL (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
NAUSEA (Gastrointestinal disorders) | 1 | 1 | 5 | 10 | 5
OESOPHAGEAL PAIN (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
STOMATITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
TOOTH LOSS (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
VOMITING (Gastrointestinal disorders) | 2 | 1 | 4 | 8 | 6
ASTHENIA (General disorders) | 0 | 0 | 0 | 1 | 3
CHEST PAIN (General disorders) | 0 | 0 | 1 | 1 | 1
CHILLS (General disorders) | 0 | 0 | 2 | 1 | 3
FACE OEDEMA (General disorders) | 0 | 0 | 1 | 0 | 0
FATIGUE (General disorders) | 0 | 0 | 6 | 7 | 8
GAIT DISTURBANCE (General disorders) | 0 | 0 | 0 | 2 | 0
INFLUENZA LIKE ILLNESS (General disorders) | 0 | 0 | 1 | 1 | 1
MALAISE (General disorders) | 0 | 0 | 0 | 1 | 1
MUCOSAL INFLAMMATION (General disorders) | 2 | 0 | 0 | 0 | 0
NON-CARDIAC CHEST PAIN (General disorders) | 0 | 1 | 0 | 0 | 0
OEDEMA (General disorders) | 0 | 0 | 2 | 1 | 1
OEDEMA PERIPHERAL (General disorders) | 0 | 1 | 2 | 2 | 1
PAIN (General disorders) | 0 | 0 | 0 | 0 | 1
PYREXIA (General disorders) | 1 | 1 | 2 | 2 | 3
SWELLING (General disorders) | 0 | 0 | 0 | 0 | 1
BRONCHITIS (Infections and infestations) | 0 | 0 | 0 | 1 | 0
CANDIDA INFECTION (Infections and infestations) | 1 | 0 | 0 | 0 | 0
CELLULITIS (Infections and infestations) | 0 | 0 | 0 | 1 | 0
CONJUNCTIVITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 1
CYSTITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 1
DIVERTICULITIS (Infections and infestations) | 0 | 0 | 1 | 0 | 0
EYE INFECTION (Infections and infestations) | 0 | 0 | 1 | 0 | 0
FUNGAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 1 | 0
LUNG INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 1
NASOPHARYNGITIS (Infections and infestations) | 0 | 0 | 0 | 1 | 0
ORAL CANDIDIASIS (Infections and infestations) | 0 | 0 | 0 | 3 | 1
PAROTITIS (Infections and infestations) | 0 | 0 | 0 | 1 | 0
PNEUMONIA (Infections and infestations) | 0 | 0 | 1 | 0 | 0
SALMONELLOSIS (Infections and infestations) | 0 | 0 | 1 | 0 | 0
SEPSIS (Infections and infestations) | 0 | 0 | 1 | 0 | 0
SINUSITIS (Infections and infestations) | 0 | 0 | 0 | 2 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 0 | 4 | 4 | 2
URINARY TRACT INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 1
VIRAL INFECTION (Infections and infestations) | 0 | 0 | 1 | 0 | 0
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 0 | 2 | 0
CONTUSION (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 2
FALL (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 1 | 2
LACERATION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
SKIN ABRASION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
TOXICITY TO VARIOUS AGENTS (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
WOUND (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 0 | 0 | 1 | 1
ASPARTATE AMINOTRANSFERASE (Investigations) | 0 | 0 | 0 | 0 | 1
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 0 | 0 | 1 | 2
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 2
BLOOD BILIRUBIN INCREASED (Investigations) | 0 | 0 | 0 | 1 | 1
BLOOD CREATININE INCREASED (Investigations) | 0 | 0 | 2 | 2 | 3
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 0 | 0 | 0 | 1 | 1
BLOOD LACTIC ACID INCREASED (Investigations) | 0 | 0 | 0 | 0 | 1
BLOOD THYROID STIMULATING HORMONE INCREASED (Investigations) | 0 | 0 | 0 | 1 | 0
ELECTROCARDIOGRAM QT PROLONGED (Investigations) | 0 | 0 | 1 | 1 | 0
GLOMERULAR FILTRATION RATE DECREASED (Investigations) | 0 | 0 | 1 | 0 | 0
HUMAN EPIDERMAL GROWTH FACTOR RECEPTOR DECREASED (Investigations) | 0 | 0 | 1 | 0 | 0
INTERNATIONAL NORMALISED RATIO DECREASED (Investigations) | 0 | 0 | 1 | 0 | 0
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 0 | 0 | 1 | 0 | 0
LYMPHOCYTE COUNT DECREASED (Investigations) | 0 | 0 | 1 | 0 | 0
NEUTROPHIL COUNT DECREASED (Investigations) | 0 | 0 | 2 | 2 | 4
NEUTROPHIL COUNT INCREASED (Investigations) | 0 | 0 | 0 | 0 | 1
PLATELET COUNT DECREASED (Investigations) | 0 | 0 | 1 | 3 | 1
PROTEIN TOTAL DECREASED (Investigations) | 0 | 0 | 1 | 0 | 1
WEIGHT DECREASED (Investigations) | 1 | 0 | 0 | 0 | 0
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 0 | 0 | 0 | 1 | 4
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 | 0 | 1 | 3 | 1
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 1 | 2 | 2 | 0
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
HYPERCHLORAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2 | 3
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 3
HYPERMAGNESAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
HYPERPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2
HYPERURICAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2 | 2
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2 | 3
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2 | 3
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 2 | 3 | 2
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 2 | 4 | 5
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 3 | 1 | 2
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 2
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3 | 2 | 1
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
JAW DISORDER (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 1
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1 | 0
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 0
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 2
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3 | 0 | 1
PAIN IN JAW (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
MELANOCYTIC NAEVUS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
AMNESIA (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
APHASIA (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
COGNITIVE DISORDER (Nervous system disorders) | 1 | 0 | 1 | 0 | 0
DEMENTIA ALZHEIMER'S TYPE (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
DEPRESSED LEVEL OF CONSCIOUSNESS (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
DIZZINESS (Nervous system disorders) | 0 | 0 | 2 | 2 | 4
DYSGEUSIA (Nervous system disorders) | 1 | 0 | 1 | 0 | 1
HEADACHE (Nervous system disorders) | 0 | 0 | 0 | 3 | 4
HYPERSOMNIA (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
HYPOAESTHESIA (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
MEMORY IMPAIRMENT (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
NEURALGIA (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
NEUROPATHY PERIPHERAL (Nervous system disorders) | 0 | 0 | 0 | 4 | 1
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 0 | 0 | 1 | 2 | 1
SEIZURE (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
SOMNOLENCE (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
SYNCOPE (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
TREMOR (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
AGITATION (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
ANXIETY (Psychiatric disorders) | 0 | 0 | 2 | 2 | 0
CONFUSIONAL STATE (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
INSOMNIA (Psychiatric disorders) | 0 | 0 | 2 | 2 | 4
MOOD ALTERED (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
MOOD SWINGS (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
RESTLESSNESS (Psychiatric disorders) | 0 | 0 | 1 | 2 | 0
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
DYSURIA (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
HAEMATURIA (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
URINARY RETENTION (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
PELVIC PAIN (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 3 | 2
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2 | 3
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0
HYPERCAPNIA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 3 | 0
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 3
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
RESPIRATORY TRACT CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 3
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0
SINUS PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
SNEEZING (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
UPPER-AIRWAY COUGH SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
BLISTER (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 1
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1
RASH (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 1
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
SKIN ULCER (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 | 0 | 0 | 0 | 1
HOT FLUSH (Vascular disorders) | 0 | 0 | 0 | 0 | 1
HYPERTENSION (Vascular disorders) | 0 | 0 | 0 | 0 | 2
HYPOTENSION (Vascular disorders) | 0 | 0 | 1 | 0 | 0
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 0 | 0 | 2 | 0 | 0
PHLEBITIS (Vascular disorders) | 0 | 0 | 0 | 1 | 0
VASCULAR RUPTURE (Vascular disorders) | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2019-07-30): https://cdn.clinicaltrials.gov/large-docs/35/NCT01999335/Prot_000.pdf
  • Statistical Analysis Plan (2016-06-21): https://cdn.clinicaltrials.gov/large-docs/35/NCT01999335/SAP_001.pdf